CLINICAL TRIAL: NCT00881647
Title: Cognitive Behavioral Treatment of Insomnia in Posttraumatic Stress Disorder
Brief Title: Treating People With Post-Traumatic Stress Disorder With Cognitive Behavioral Therapy for Insomnia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R34MH077667 (NIH); R34MH077667 (NIH); DATR AD-TS
Record Dates: First submitted 2009-04-14; First posted 2009-04-15 (Estimated); Results first posted 2014-02-21 (Estimated); Last update posted 2014-03-17 (Estimated); Status verified 2014-02

CONDITIONS: Post-Traumatic Stress Disorder
Keywords: PTSD; Insomnia Disorder; Insomnia; CBT
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Participants will receive an 8-week course of cognitive behavioral therapy for insomnia.
  Interventions: Other: Cognitive Behavioral Treatment for Insomnia (CBT-I)
- 2 (No Intervention): Participants will be placed on a waitlist for 8 weeks.

INTERVENTIONS:
Other: Cognitive Behavioral Treatment for Insomnia (CBT-I) — CBT-I includes strategies and instructions targeted toward improving the quality of sleep and resolving problems falling and staying asleep
  Arms: 1

SUMMARY:
This study will test the effectiveness of cognitive behavioral therapy for insomnia in treating sleep disturbances in people with post-traumatic stress disorder.

DETAILED DESCRIPTION:
Cognitive behavioral therapy to treat insomnia (CBT-I) was developed for people with primary insomnia but has been successfully used to treat insomnia in people with other disorders. Insomnia is the most commonly reported complaint of patients receiving treatment for post-traumatic stress disorder (PTSD). Medications are not effective in treating insomnia in people with PTSD, and behavioral treatments, like CBT-I, have not yet been proven effective in these cases. This study will test the effectiveness of CBT-I in alleviating insomnia in people with PTSD.

Participation in this study will last 10 months. At study entry, participants will complete a series of eligibility assessments, including a clinical interview, a medical screening, a urine screening for drugs of abuse, a blood test, and a pregnancy test. Then, over 1 week, participants will complete baseline assessments of sleep behaviors. The assessments will include the following: filling out a set of questionnaires about health, mood, sleeping patterns, possible life trauma, and PTSD; filling out a sleep diary every morning to record time slept, times woken up, nightmares, and quality of sleep; wearing a wristwatch-like device, called an Actigraph, that records activity level during wakefulness and sleep; completing a 5-minute psychomotor vigilance task twice a day on a personal digital assistant (PDA); wearing a sensor connected to the finger that detects sleep apnea, called an Oximeter, 1 night while sleeping; and, during the last 2 nights of sleep assessment, having a sleep recorder connected to one's head to measure different stages of sleep.

After the week of sleep assessments, participants will be randomly assigned to one of two groups: the CBT-I group or the waitlist group. Participants in the CBT-I group will complete eight weekly therapy sessions targeted at improving quality of sleep and resolving problems with falling and staying asleep. Participants in the waitlist group will not be offered CBT-I treatment until after 8 weeks. During these 8 weeks, all participants will continue to keep a sleep diary, continue wearing the Actigraph, and, in the fourth week, be asked to fill out a questionnaire booklet with similar questions to those completed in the eligibility screening. After 8 weeks, participants will repeat all the sleep assessments performed at baseline. They will also undergo a clinical interview to assess the severity of PTSD symptoms and sleep problems. After the second set of sleep assessments, the waitlist group will be offered CBT-I, and the CBT-I group will complete 6- and 12-month follow-up assessments. These follow-up assessments will involve repeating both the sleep assessments and the clinical interview performed after the 8-week intervention.

ELIGIBILITY:
Inclusion Criteria:

* Chronic PTSD for at least 3 months
* Currently on first line treatment for PTSD, defined as selective serotonin reuptake inhibitor (SSRI) therapy, for at least 6 months
* Persistent residual insomnia

Exclusion Criteria:

* Conditions or substances that may be associated with comorbid insomnia independent of PTSD

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2008-11; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas C. Neylan, MD, Principal Investigator — University of California, San Francisco/VA Medical Center, San Francisco
Locations (1):
- VA Medical Center, San Francisco, San Francisco, California, United States

REFERENCES:
- [Derived] Kanady JC, Talbot LS, Maguen S, Straus LD, Richards A, Ruoff L, Metzler TJ, Neylan TC. Cognitive Behavioral Therapy for Insomnia Reduces Fear of Sleep in Individuals With Posttraumatic Stress Disorder. J Clin Sleep Med. 2018 Jul 15;14(7):1193-1203. doi: 10.5664/jcsm.7224. PMID 29991428
- [Derived] Talbot LS, Maguen S, Metzler TJ, Schmitz M, McCaslin SE, Richards A, Perlis ML, Posner DA, Weiss B, Ruoff L, Varbel J, Neylan TC. Cognitive behavioral therapy for insomnia in posttraumatic stress disorder: a randomized controlled trial. Sleep. 2014 Feb 1;37(2):327-41. doi: 10.5665/sleep.3408. PMID 24497661
- See also: More information about the Stress & Health Research Program — http://www.stressandhealthresearch.com

RESULTS

PARTICIPANT FLOW:
Groups:
- CBT-I: 8-week course of Cognitive Behavioral Treatment for Insomnia (CBT-I): CBT-I includes strategies and instructions targeted toward improving the quality of sleep and resolving problems falling and staying asleep
- Waitlist: Participants placed on a waitlist for 8 weeks.
Period: Overall Study
Arm/Group | CBT-I | Waitlist
Started | 29 | 16
Completed | 27 | 15
Not Completed | 2 | 1

BASELINE CHARACTERISTICS:
Population: per protocol
Groups:
- Total: Total of all reporting groups
Arm/Group | CBT-I | Waitlist | Total
Number analyzed (Participants) | 29 | 16 | 45
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.1 (10.4) | 37.3 (11.0) | 37.2 (10.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 9 | 31
  Male | 7 | 7 | 14
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 3 | 2 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 5 | 1 | 6
  White | 20 | 12 | 32
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 1 | 2
Region of Enrollment [Number; unit: participants]
  United States | 29 | 16 | 45
Marital Status [Number; unit: participants]
  Single | 20 | 10 | 30
  Married/Partnered | 6 | 2 | 8
  Divorced | 3 | 3 | 6
  Separated | 0 | 1 | 1
Veteran Status [Number; unit: participants]
  Veteran | 3 | 6 | 9
  Not veteran | 26 | 10 | 36
PTSD Duration [Mean (Standard Deviation); unit: years] | 20.4 (13.6) | 15.0 (13.8) | 18.5 (2.1)
Current Depression [Number; unit: participants] — Depression symptoms were assessed using the Beck Depression Inventory
  participants
    Depressed | 5 | 4 | 9
    Not depressed | 24 | 12 | 36
Using psychotropic medication [Number; unit: participants]
  Using psychotropic medication | 11 | 7 | 18
  Not using psychotropic medication | 18 | 9 | 27

OUTCOME MEASURES:

1. Primary Outcome: Sleep Latency (SL)
Description: In a self-report sleep diary, participants were asked to report the length of time it takes from lying down for the night until sleep onset. This outcome consists of the posttreatment (CBT-I) or post-waitlist diary entry; In other words, each of the values below was measured at 8 weeks.
Time Frame: After 8 weeks of study participation
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | CBT-I | Waitlist
Number analyzed (Participants) | 27 | 15
minutes | 14.27 (2.27) | 44.31 (11.72)

2. Primary Outcome: Minutes of Wake After Sleep Onset (WASO)
Description: WASO was the sum of wake time during sleep as recorded in a self-report sleep diary, and as measured in epochs (30 seconds of polysomnography [PSG]) recording) after the onset of persistent sleep and prior to final awakening and wake time after sleep (the number of epochs after the final awakening until the end of PSG recording [i.e. awake epoch immediately prior to the end of the recording]). This outcome consists of posttreatment (CBT-I) or post-waitlist diary entries and polysomnography data; In other words, each of the values below was measured at 8 weeks.
Time Frame: After 8 weeks of study participation
Population: per protocol
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | CBT-I | Waitlist
Number analyzed (Participants) | 27 | 15
Minutes
  WASO by self report | 13.82 (2.03) | 47.25 (11.45)
  WASO by PSG | 39.25 (7.73) | 57.63 (18.28)

3. Primary Outcome: Sleep Efficiency (SE)
Description: SE, as determined by polysomnography (PSG) and by self-reported sleep diary, was the total sleep time (TST) divided by the time in bed, multiplied by 100. This outcome consists of posttreatment (CBT-I) or post-waitlist diary entries and polysomnography data; In other words, each of the values below was measured at 8 weeks.
Time Frame: After 8 weeks of study participation
Measure: Mean (Standard Deviation); unit: percentage of time
Arm/Group | CBT-I | Waitlist
Number analyzed (Participants) | 27 | 15
percentage of time
  SE by self-report | 93.72 (0.93) | 81.77 (2.47)
  SE by PSG | 91.35 (1.91) | 88.14 (3.59)

ADVERSE EVENTS:
Time Frame: 8 weeks
Arm/Group | CBT-I | Waitlist
Serious Adverse Events (participants affected / at risk) | 0/29 | 0/16
Other Adverse Events (participants affected / at risk) | 0/29 | 0/16

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes